CLINICAL TRIAL: NCT07026435
Title: Comparison of Lesion Sterilization and Tissue Repair Technique With Conventional Pulpectomy in the Treatment of Pulpal Lesions in Primary Molars in Children
Brief Title: Comparison of LSTR and Pulpectomy in Primary Molars of Pediatric Patients (LSTR-PULP)
Acronym: LSTR-PULP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: taymour abuawwad (Other)
Responsible Party: Sponsor-Investigator, taymour abuawwad, PhD Candidate in Pediatric Dentistry, Ataturk University
Organization: Ataturk University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/477; TDK-2024-14564 (Other: Ataturk University Scientific Research Projects Unit (BAP))
Record Dates: First submitted 2025-05-19; First posted 2025-06-18 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Pulpal Necrosis; Dental Caries; Periapical Periodontitis; Pediatric Dentistry; Primary Tooth Pulpectomy
Keywords: LSTR; Pulpectomy; Primary teeth; Triple antibiotic paste
MeSH Terms: conditions — Dental Pulp Necrosis; Dental Caries; Periapical Periodontitis | interventions — Pulpectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSTR Group (Experimental): Children will receive the LSTR (Lesion Sterilization and Tissue Repair) procedure, which includes applying a mixture of ciprofloxacin and metronidazole with iodoform-calcium hydroxide paste to the pulp chamber without canal instrumentation. Restoration will be done using a stainless steel crown or compomer.
  Interventions: Procedure: LSTR
- Pulpectomy Group (Active Comparator): Children will receive conventional pulpectomy involving mechanical canal instrumentation and obturation with iodoform-calcium hydroxide paste. Restoration will be completed with a stainless steel crown or compomer based on clinical conditions.
  Interventions: Procedure: Pulpectomy

INTERVENTIONS:
Procedure: LSTR — Lesion Sterilization and Tissue Repair (LSTR) is a minimally invasive pulp therapy using ciprofloxacin and metronidazole mixed with iodoform-calcium hydroxide, without canal instrumentation. The access cavity is sealed and restored with SSC or compomer.
  Arms: LSTR Group
Procedure: Pulpectomy — Pulpectomy includes mechanical canal preparation, irrigation, and obturation using iodoform-calcium hydroxide paste, followed by final restoration with stainless steel crown or compomer.
  Arms: Pulpectomy Group

SUMMARY:
This study aims to compare the effectiveness of Lesion Sterilization and Tissue Repair (LSTR) with conventional pulpectomy in treating pulpal lesions in primary molars of pediatric patients aged 4 to 10 years. LSTR is a minimally invasive method that uses antibiotic paste to disinfect infected tissue without full canal instrumentation. Children participating in this study will receive either the LSTR technique or standard pulpectomy, and the clinical and radiographic success of both treatments will be evaluated over a 12-month period. The goal is to determine whether LSTR is a safe and effective alternative to pulpectomy in primary teeth.

DETAILED DESCRIPTION:
This is a prospective, clinical trial conducted at Atatürk University, Department of Pediatric Dentistry. The study compares two endodontic treatment methods for primary molars with pulpal lesions in children aged 4 to 10 years. A total of 108 primary molars will be assigned to two groups: the experimental group receiving Lesion Sterilization and Tissue Repair (LSTR) and the control group receiving conventional pulpectomy. The LSTR group will be treated with a combination of ciprofloxacin and metronidazole antibiotics mixed with iodoform-calcium hydroxide paste, while the pulpectomy group will receive standard chemomechanical canal debridement and obturation with iodoform-calcium hydroxide paste. Each treatment will be followed by restoration using either compomer or stainless steel crown, depending on patient cooperation and clinical setting. Patients will be followed up clinically at 3, 6, and 12 months and radiographically at 6 and 12 months. Treatment success will be evaluated based on the resolution of clinical symptoms and radiographic healing, using the Periapical Index (PAI) and observation of root resorption patterns. The primary objective is to assess whether the LSTR technique achieves similar or superior success rates compared to pulpectomy in terms of both clinical outcomes and radiographic healing.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 10 years.
* Presence of at least one primary molar with pulpal involvement requiring endodontic treatment.
* Good general health without systemic conditions.
* Signed informed consent from parent or legal guardian.

Exclusion Criteria:

* Children with systemic diseases or immune-compromising conditions.
* Known allergies to any of the materials or antibiotics used in the study.
* Uncooperative behavior preventing dental treatment under normal clinical conditions.
* Teeth with non-restorable crown structure or excessive root resorption.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-10-08 (Estimated)

PRIMARY OUTCOMES:
Clinical Success Rate of Treated Primary Molars | At 3, 6, and 12 months post-treatment
  Clinical success is defined as absence of pain, swelling, sinus tract, and pathological mobility assessed through standardized clinical examination by a pediatric dentist.

SECONDARY OUTCOMES:
Radiographic Healing Rate of Treated Primary Molars | At 6 and 12 months post-treatment
  Radiographic healing is defined as the resolution of periapical or furcal radiolucency and the absence of pathological root resorption. This will be assessed using the Periapical Index (PAI) scoring system (scale range 1 to 5, where lower scores indicate better healing) by two calibrated evaluators using digital radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Sera DERELİOĞLU, DDS, PhD, Principal Investigator — Ataturk University
Locations (1):
- Atatürk University Faculty of Dentistry, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT07026435/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT07026435/ICF_001.pdf